CLINICAL TRIAL: NCT04950010
Title: Enhancing Cognitive and Cardiovascular Function in Breast Cancer Survivors Through High-intensity Interval Training
Brief Title: High-intensity Exercise After Treatment
Acronym: HEAT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Original PI moved to a new institution
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 0439-21-FB; 1U54GM115458 (NIH)
Record Dates: First submitted 2021-06-14; First posted 2021-07-02 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer; Breast Neoplasm Female
Keywords: breast cancer; physical activity; cognitive function; exercise; cardiovascular function
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-Intensity Interval Training (HIIT) (Experimental): Breast cancer survivors randomized to HIIT will participate in a high-intensity interval training program for 8 weeks.
  Interventions: Behavioral: High-Intensity Interval Training
- Moderate-Intensity Exercise (MOD) (Active Comparator): Breast cancer survivors randomized to MOD will participate in a moderate-intensity aerobic exercise program for 8 weeks.
  Interventions: Behavioral: Moderate-Intensity Exercise
- Usual Care (UC) (No Intervention): Individuals randomized to UC will be instructed to continue standard cancer care and engage in habitual lifestyle behaviors.

INTERVENTIONS:
Behavioral: High-Intensity Interval Training — HIIT is a type of training in which short periods of high-intensity anaerobic exercise (1-4 minutes at 80-95% of VO2peak) are alternated with less intense aerobic recovery periods (1-3 minutes at 50-60% VO2peak). Individually-tailored exercise prescriptions will be developed based upon each participant's baseline maximal graded exercise test (heart rate corresponding with %VO2 peak) and symptom limitation. Sessions will be progressive in nature such that the volume of exercise (i.e., number and intensity of intervals) increases across weeks. Intervals will progress from a heart rate corresponding with 75% VO2peak in Week 1 to 90-95% VO2peak in Weeks 5-8. Sessions will be ~30 minutes in length. Indoor cycling is the primary mode of exercise.
  Arms: High-Intensity Interval Training (HIIT)
Behavioral: Moderate-Intensity Exercise — Individually-tailored exercise prescriptions will be developed based upon each participant's baseline maximal graded exercise test (heart rate corresponding with %VO2 peak) and symptom limitation. Sessions will be progressive in nature such that the volume of exercise increases across weeks. Indoor cycling is the primary mode of exercise. Sessions will include moderate-intensity cycling that progresses from a heart rate corresponding with 55-60% VO2peak for 30 minutes in Week 1 to 65-70% VO2peak for 45-50 minutes in Weeks 5-8.
  Arms: Moderate-Intensity Exercise (MOD)

SUMMARY:
This pilot study tests the feasibility and preliminary efficacy of an 8-week, 3-arm pilot exercise trial in which 45 breast cancer survivors will be randomized to high-intensity interval training (HIIT; n=15), moderate-intensity aerobic training (MOD; n=15), or Usual Care (UC; n=15).

DETAILED DESCRIPTION:
Aim 1: Determine the feasibility and acceptability of an 8-week high-intensity interval training (HIIT) program compared with a standard moderate-intensity aerobic training (MOD) program in 45 breast cancer survivors prescribed aromatase inhibitors.

Aim 2: Calculate effect sizes associated with the 8-week HIIT program, compared with MOD and Usual Care (UC), on cognitive and cardiovascular functions in 45 breast cancer survivors.

Eligible individuals will be women diagnosed with Stages I-IIIa breast cancer, have completed primary treatment (i.e., surgery, chemotherapy, and/or radiation therapy), and currently prescribed an aromatase inhibitor. The specific aims are: 1) Determine the feasibility and acceptability of an 8-week high-intensity interval training (HIIT) program compared with a standard moderate-intensity (MOD) program; and 2) Calculate effect sizes associated with the 8-week HIIT program, compared with MOD and usual care (UC), on cognitive and cardiovascular functions. Cognitive function is operationalized as performance on executive function and working memory tasks. Cardiovascular function is operationalized as exercise capacity (VO2peak, heart rate recovery), resting function (heart rate, blood pressure), and cardiovascular structure/function (arterial stiffness, arterial wall thickness, endothelial function). Associations between change in cardiovascular outcomes and change in cognitive outcomes across the intervention period will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* Adult female (aged 19 or older)
* First, primary diagnosis of Stage I-IIIa breast cancer
* Hormone receptor positive (ER+ and/or PR+) diagnosis
* Human epidermal growth factor receptor 2 negative (HER2-) diagnosis
* Completed primary adjuvant treatment (i.e., surgery, chemotherapy, and/or radiation therapy)
* Currently prescribed an aromatase inhibitor
* No evidence of possible cognitive impairment as assessed using the Telephone Interview of Cognitive Status (TICS-M; score >21)
* Sedentary except for casual lifestyle recreation. This is defined as self-reporting 20+ minutes of exercise physical activity on 2 or fewer days per week within the previous six months.
* Receive physician's clearance to participate in an exercise program
* Agree to be randomized
* Fully vaccinated for COVID-19 ≥2 weeks prior to participation
* Provide written informed consent to participate in study

Exclusion Criteria:

* Males.
* Stage 0 breast cancer diagnosis or metastatic disease
* Currently receiving chemotherapy or radiation therapy for any cancer
* Scheduled to receive breast surgery (e.g., mastectomy, reconstructive surgery) during the study period
* Second cancer diagnosis (excluding non-invasive skin cancers; including breast cancer recurrence)
* Self-report an 20+ minutes of exercise physical activity on 3+ days per week for the previous 6 months
* Pregnant or plan to become pregnant during study period.
* Is not cleared to participate in exercise by a physician.
* Enrolled in another physical activity program
* Unable to cycle on a stationary bike
* Unwilling to complete study requirements
* History of stroke, transient ischemic attack, other neurological disorders, or brain surgery involving tissue removal
* Clinically significant TICS-M score (<21) during baseline procedures
* Not fully vaccinated for COVID-19

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Participation Rate | Baseline
  Sample size / [1-(#ineligible/# exposed to recruitment)*(#exposed to recruitment)]
Adherence to the exercise programs | post-intervention (Week 9)
  average number of exercise sessions (out of 24) attended
Compliance of the exercise programs | post-intervention
  average number of exercise sessions (out of 24) in which the prescribed exercise duration and intensity are achieved
Acceptability of the exercise programs | post-intervention
  satisfaction with the exercise program as measured by a satisfaction survey. Survey uses a 5-point Likert-type scale. Satisfaction for each item is defined as reporting 4-5 on the scale (i.e., somewhat agree or completely agree).
Change in executive function processing | Baseline, post-intervention (Week 9)
  Change in completion time on Trails B task, with higher values indicating lower executive function.
Change in cognitive flexibility | Baseline, post-intervention (Week 9)
  Change in reaction time on Task-switch task, with higher values indicating lower cognitive flexibility
Change in spatial working memory reaction time | Baseline, post-intervention (Week 9)
  Change in reaction time on spatial working memory task, with faster reaction times indicating better spatial working memory

SECONDARY OUTCOMES:
Change in Cardiorespiratory Fitness | Baseline, post-intervention (Week 9)
  Change in Peak VO2 as measured by a modified Balke treadmill graded exercise test protocol.
Carotid arterial wall thickness | Baseline, post-intervention (Week 9)
  will be estimated from vascular ultrasound and expressed as average and maximum mm
Endothelial function | Baseline, post-intervention (Week 9)
  estimated from brachial artery flow mediated dilation and expressed as percent change in brachial artery diameter relative to baseline diameter

CONTACTS AND LOCATIONS:
Overall Officials: Diane Ehlers, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Although the final dataset will not include identifying information, there is still a possibility of deductive disclosure of identity. Therefore, data will not be shared via an NIH or approved public repository; however, we will share de-identified data as required for publication in scientific journals and with outside collaborators and scientists upon request.
Supporting Information: Study Protocol
Time Frame: Data will be shared via scientific journals at the time of publication and with outside collaborators before publication.
Access Criteria: We will make data available to researchers who agree to use the data only for research purposes, protect the data using secure computer technologies, and destroy the data after relevant analyses are completed and manuscripts published.